CLINICAL TRIAL: NCT00838136
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Lamotrigine 25 mg Chewable Dispersible Tablets and Lamictal® 25 mg Chewable Dispersible Tablets in Healthy Subjects Under Fed Conditions
Brief Title: Lamotrigine 25 mg Chewable Tablets, Non-Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01304
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (Experimental): Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in first period followed by Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in second period
  Interventions: Drug: Lamotrigine 25 mg Chewable Tablets
- Lamictal® (Active Comparator): Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in first period followed by Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in second period
  Interventions: Drug: Lamictal® 25 mg Chewable Tablets

INTERVENTIONS:
Drug: Lamotrigine 25 mg Chewable Tablets — 2 x 25 mg, single-dose fed
  Arms: Lamotrigine
Drug: Lamictal® 25 mg Chewable Tablets — 2 x 25 mg, single-dose fed
  Arms: Lamictal®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of lamotrigine 25 mg chewable dispersible tablets (test) versus Lamictal® (reference) administered as 2 x 25 mg chewable dispersible tablets under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Female subjects will be post-menopausal or surgically sterilized.
* Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Subjects with a history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm) at screening.
* Subjects with BMI ≥ 30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit - 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PVP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* History of allergic reactions to lamotrigine.
* Use of any drugs known to induce or inhibit drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine, valproic acid), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Subjects who have dentures or braces.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follow: less than 300 mL of whole blood within 30 days; 300 mL to 500 mL of whole blood within 45 days; more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within 90 days preceding study drug administration.
* Female subjects: breast-feeding subjects.
* Female subjects: positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-02; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine (Test) First: Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in first period followed by Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in second period
- Lamictal® (Reference) First: Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in first period followed by Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 14 | 16 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 13 | 14 | 27
  American Hispanic | 3 | 0 | 3
  Black | 0 | 1 | 1
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lamotrigine: Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in either period
- Lamictal®: Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in either period
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 31 | 31
ng/mL | 612.45 (66.77) | 604.85 (67.94)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 101.23, 90% CI [99.88 to 102.60] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 31 | 31
ng*h/mL | 33783.02 (11635.51) | 32950.62 (9855.72)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 101.87, 90% CI [99.18 to 104.63] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 31 | 31
ng*h/mL | 28968.25 (6132.36) | 28687.23 (5638.21)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 100.76, 90% CI [98.60 to 102.97] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.